CLINICAL TRIAL: NCT00064922
Title: Incentive Programs for Female Substance Abusers Who Smoke
Brief Title: Incentive Programs for Female Substance Abusers Who Smoke - 3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-13638-3; R01-13638-3
Record Dates: First submitted 2003-07-15; First posted 2003-07-16 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-05

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to examine the effects of incentive programs for the treatment of nicotine dependence in women who have problems with substance dependence.

DETAILED DESCRIPTION:
This study will determine the influence of voucher-based CM on reducing smoking (and other drug) use during pregnancy or in post-partum women with children under 1 year of age living with them, or in non-pregnant females who smoke. We are targeting smoking cessation since cigarette use is so prevalent in our service. We will compare a control group to two different voucher-based contingent-reinforcement procedures: one that targets smoking abstinence alone vs. one that offers additional incentives for negative BAL and urinalysis results.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and or post-partum with at least one child under 1 year old living with them, or non-pregnant, non-post-partum females or previous participant in this study protocol
* Nicotine Dependent as confirmed by DSM-IV checklist
* Current cigarette smoker
* Breath CO reading of at least 8 ppm at the time of the initial study screening
* Current client with the Shields for Families (Shields) treatment programs

Exclusion Criteria:

* Non-smoker

Ages: 15 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2002-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — Los Angeles Treatment Research Center
Locations (1):
- Shields for Families, Inc., Los Angeles, California, United States